CLINICAL TRIAL: NCT01853072
Title: Randomized, Double-Masked, Vehicle Controlled, Clinical Evaluation To Assess The Safety And Efficacy Of Nepafenac Ophthalmic Suspension, 0.3% For Improvement In Clinical Outcomes Among Diabetic Subjects Following Cataract Surgery
Brief Title: Nepafenac Once Daily for Macular Edema - Study 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-12-067
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-06

CONDITIONS: Non-Proliferative Diabetic Retinopathy; Cataract
Keywords: Diabetes Type I; Diabetes Type II; non-proliferative diabetic retinopathy; macular edema; Cataract
MeSH Terms: conditions — Cataract; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Macular Edema | interventions — nepafenac; prednisolone acetate; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nepafenac (Experimental): With prednisolone acetate standard of care, Nepafenac Ophthalmic Suspension, 0.3%, 1 drop instilled in the operative eye 1 day prior to surgery, continuing on the day of surgery, and for 90 days following surgery. An additional 1 drop will be administered 30 to 120 minutes prior to surgery.
  Interventions: Drug: Nepafenac Ophthalmic Suspension, 0.3%; Drug: Prednisolone acetate
- Vehicle (Placebo Comparator): With prednisolone acetate standard of care, Nepafenac vehicle, 1 drop instilled in the operative eye 1 day prior to surgery, continuing on the day of surgery, and for 90 days following surgery. An additional 1 drop will be administered 30 to 120 minutes prior to surgery.
  Interventions: Other: Nepafenac vehicle; Drug: Prednisolone acetate

INTERVENTIONS:
Drug: Nepafenac Ophthalmic Suspension, 0.3% — Test intervention
  Other Names: Nepafenac
  Arms: Nepafenac
Other: Nepafenac vehicle — Inactive ingredients used as placebo comparator
  Arms: Vehicle
Drug: Prednisolone acetate — 1 drop instilled in the operative eye 4 times daily beginning post-operatively on the day of surgery for the first 2 weeks, followed by 2 times daily for the next 2 weeks
  Other Names: Omnipred™; Prednisolone acetate ophthalmic suspension

SUMMARY:
The purpose of this study is to demonstrate superiority of Nepafenac Ophthalmic Suspension, 0.3% dosed once daily relative to Nepafenac Vehicle based upon clinical outcomes among diabetic subjects following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planned cataract extraction by phacoemulsification with implantation of a posterior chamber intraocular lens;
* History of Type 1 or 2 diabetes and non-proliferative diabetic retinopathy (NPDR) (mild, moderate, or severe) in the study eye;
* Best corrected visual acuity (BCVA) of 73 letters or worse in the study eye with expectation of improvement after surgery;
* Understand and sign an informed consent document;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Pre-existing macular edema in the study eye;
* History in the study eye of retinal detachment, wet age-related macular degeneration, chronic or recurrent inflammatory eye disease, or prior procedures;
* Planned cataract surgery in the fellow eye after randomization and prior to the Day 90 postoperative study visit or through study exit;
* Planned multiple procedures for the study eye during the cataract/intraocular lens implantation surgery;
* Use of exclusionary medications, including nonsteroidal anti-inflammatory drugs (NSAIDs) and steroids, as specified in protocol.
* Participation in any other clinical study within 30 days of the screening visit;
* Females of childbearing potential who are breast feeding, have a positive urine pregnancy test at screening, are not willing to undergo a urine pregnancy test upon entering or exiting the study, intend to become pregnant during the study, or do not agree to use adequate birth control methods for the duration of the study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 881 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Lead GCRA, Pharma, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 66 investigational centers located in the U.S., Latin America, and the Caribbean.
Pre-assignment Details: Of the 881 participants enrolled, 253 were exited as screen failures and 13 were discontinued prior to randomization. This reporting group includes all randomized participants (615).
Groups:
- Nepafenac: Nepafenac Ophthalmic Suspension, 0.3%
- Vehicle: Nepafenac Ophthalmic Suspension Vehicle
Period: Overall Study
Arm/Group | Nepafenac | Vehicle
Started | 308 | 307
Randomized | 308 | 307
Treated (Safety Analysis Set) | 301 | 302
Full Analysis Set | 298 | 300
Completed | 296 | 286
Not Completed | 12 | 21
Not completed — Adverse event prior to treatment | 0 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Death | 1 | 4
Not completed — Lost to Follow-up | 0 | 3
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Reason not specified | 9 | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set, defined as including all randomized participants who completed implant surgery and had at least one on-therapy postsurgical visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nepafenac | Vehicle | Total
Number analyzed (Participants) | 298 | 300 | 598
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (8.5) | 66.8 (8.3) | 66.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 166 | 324
  Male | 140 | 134 | 274

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best-corrected Visual Acuity (BCVA) Improvement of ≥ 15 Letters From Preoperative Baseline to Day 14 and Maintained Through Day 90
Description: BCVA (with spectacles or other visual corrective devices) was reported in letters read correctly, using the Early Treatment Diabetic Retinopathy Study (ETDRS) test of 70 letters. Improvement of BCVA was defined as an increase (gain) in the number of letters read, compared to the baseline assessment. One eye (study eye) contributed to the analysis.
Time Frame: Baseline to Day 14, and maintained through Day 90
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 298 | 300
Percentage of participants | 61.7 | 43.0
Statistical Analysis 1: Comparison: Nepafenac vs Vehicle; This endpoint was considered primary for United States (US) registration and secondary for European Union (EU) registration; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.1, 95% CI 2-sided [1.5 to 3.0], Standard Error of Mean 0.4 — Parameter dispersion is the standard error for the odds ratio

2. Primary Outcome: Percentage of Participants Who Develop Macular Edema Within 90 Days Following Cataract Surgery (Day 0)
Description: Macular edema was defined as ≥ 30% Increase from pre-operative baseline in central subfield macular thickness, as measured with Spectral Domain Ocular Coherence Tomography (SD-OCT). One eye (study eye) contributed to the analysis.
Time Frame: Day 0 to Day 90
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 298 | 300
Percentage of participants | 2.3 | 17.3
Statistical Analysis 1: Comparison: Nepafenac vs Vehicle; This endpoint was considered primary for EU registration and secondary for US registration; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.1, 95% CI 2-sided [0.1 to 0.3], Standard Error of Mean 0.1 — Parameter dispersion is the standard error for the odds ratio

3. Secondary Outcome: Percentage of Participants With BCVA Improvement of ≥ 15 Letters From Preoperative Baseline to Day 90
Time Frame: Baseline to Day 90
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 298 | 300
Percentage of participants | 77.2 | 67.7

4. Secondary Outcome: Percentage of Participants With BCVA Improvement of ≥ 15 Letters From Preoperative Baseline to Day 60
Time Frame: Baseline to Day 60
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 298 | 300
Percentage of participants | 76.2 | 64.7

5. Secondary Outcome: Percentage of Participants With a > 5-letter Loss in BCVA From Day 7 to Any Visit [Time Frame: Day 7 up to Any Visit]
Time Frame: Day 7 up to any visit through Day 90
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 298 | 300
percentage of participants | 15.4 | 27.3

6. Secondary Outcome: Percentage of Participants With With a > 10-letter Loss in BCVA From Day 7 to Any Visit
Time Frame: Day 7 up to any visit through Day 90
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 298 | 300
percentage of participants | 9.1 | 15.3

ADVERSE EVENTS:
Time Frame: Reporting of adverse events (AEs) began once informed consent was obtained from the subject and continued through Day 90 (or Day 120, if unresolved macular edema present at Day 90). Ocular AEs are presented for both study eye and non-study eye combined.
Description: An AE was defined as any untoward medical occurrence in a subject after signing the informed consent document. AEs were reported as pretreatment, treatment-emergent, and posttreatment. Reports of AEs were obtained through solicited and spontaneous comments from the participants.
Groups:
- Pretreatment: All participants who consented to participate in the study prior to the initiation of study treatment
- Nepafenac: All participants treated with Nepafenac during the course of study treatment
- Vehicle: All participants treated with NepafenacVehicle during the course of study treatment
- Posttreatment: All participants after cessation of study treatment up to study exit
Arm/Group | Pretreatment | Nepafenac | Vehicle | Posttreatment
Serious Adverse Events (participants affected / at risk) | 14/881 | 13/301 | 14/302 | 9/603
Other Adverse Events (participants affected / at risk) | 0/881 | 0/301 | 0/302 | 0/603
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=881) | Nepafenac (N=301) | Vehicle (N=302) | Posttreatment (N=603)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 3 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pericolic abscess (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Retroperitoneal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arteriogram (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.